CLINICAL TRIAL: NCT03215225
Title: Long-term Evaluation of Endodontic Root Canal Treatments: Complication, Factors Affecting Failure, New Disease and Success
Brief Title: Endodontic Root-canal Treatments Evaluated After Long-term Time
Acronym: ENDOBO20
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Carlo Prati, Full time Ordinary Professor, University of Bologna
Other Study IDs: Endo master treatment
Record Dates: First submitted 2017-07-09; First posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Root Canal Treatment; Endodontic Disease
Keywords: Endodontology; Endodontics
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Root canal treatment
  Interventions: Procedure: Root canal orthograde treatment

INTERVENTIONS:
Procedure: Root canal orthograde treatment

SUMMARY:
The aim of the study was to evaluate the root canal treatments performed from 1989 to 1995. Type of complication, success, new endodontic diseases and number of success were reported. Mean clinical parameters were clinical symptoms and presence/absence of apical radiolucency.

DETAILED DESCRIPTION:
See previous papers (Pirani et al., Odontology, 2015)

ELIGIBILITY:
Inclusion Criteria:

Patients affected by endodontic disease and able to attend a recall hygien program

Exclusion Criteria:

* Sistemic disease Cancer Inability to attend a recall hygien program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Similar geographic provenience
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 1989-12-01 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Health Patients | 2 years
  patients with periapical disease and/or pulpal disease

IPD SHARING:
Plan to Share IPD: No